CLINICAL TRIAL: NCT02737163
Title: Inadvertent Cerebral Spinal Fluid Valve Reprogramming: Prevalence and the Correlation With Signs, Symptoms, Radiographic Changes and the Exposure to Magnetic Fields.
Brief Title: Strata Programmable CSF Shunt Valve Study
Status: Terminated | Type: Observational
Why Stopped: Terminated early due to sufficient data acquired to meet our study objectives
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00093490
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Hydrocephalus
Keywords: Programmable shunts; Strata valve
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The treatment of hydrocephalus is the most time consuming, and arguably the most important role of the pediatric neurosurgical service at most children's' hospitals. Despite many technological advances, cerebral spinal fluid (CSF) shunting procedures remain the mainstay of hydrocephalus treatment. While often lifesaving, CSF shunting procedures are associated with high complication rates and account for a disproportionate share of health care expenditures and morbidity.

Programmable CSF shunt valves, through which CSF flow and pressure can be adjusted by quick and painless transcutaneous reprogramming, have been implanted for more than 15 years in the developed world. Reprogramming these valves relies on rotational magnetic forces, which are applied by neurosurgeons and neurosurgical advanced practice providers. Inadvertent reprogramming (IR) can occur when patients with these valves are exposed to magnetic fields in the environment, which may lead to serious symptoms that may require urgent reprogramming and/or surgery.

The concurrent proliferation of magnetically sensitive programmable CSF shunt valves and household items that generate substantial magnetic fields has caused concern among patients, parents and providers about the potential consequences of inadvertent valve reprogramming. This growing concern led the FDA to issue a warning to individuals with programmable valves in 2014, which deemed the programmable valves safe for use but vulnerable to IR when household devices such as tablets or cell phones are placed within 2 inches of the valve. The FDA recommended further study, stating that no systematic evaluation had been performed regarding the prevalence of accidental valve adjustments.

By evaluating each of the patients with magnetically susceptible CSF shunt valves, during each of the routine points of contact with the service, investigators aim to define the prevalence of inadvertent shunt reprogramming, to correlate with the presence and absence of symptoms and radiographic changes, and to evaluate the risk of inadvertent shunt reprogramming based on exposure to common environmental items.

DETAILED DESCRIPTION:
Investigators intend to evaluate all patients 21 years old and younger with magnetically susceptible CSF shunts, specifically those with Strata (Medtronic, Dublin) valves implanted. All evaluations will be performed during routine patient care in the hospital, the emergency department and in the outpatient facilities. Valve settings will be checked transcutaneously in the standard manner, before and after any MRI studies.

Evaluating IR and making correlations between exposure to MRI or environmental magnets and symptoms and radiographic changes (when available) will require the patient or family to complete a brief questionnaire. It will then require the study team and delegated providers to check the valve setting before and after MRI, and to gather clinical information from the medical record and from the current clinical evaluation.

Each patient's initial enrollment will require the acquisition of an informed consent, which will cover all future evaluations of IR during the three year study period for that patient. However, every time a patient enrolled in the study encounters the neurosurgical service, all study steps will be performed, including the valve check before and after MRI, the participant's completion of the questionnaire, and the research staff's completion of the data sheets.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21 years of age and younger
* With Strata valve CSF shunts
* Who are being evaluated by the All Children's Hospital (ACH) neurosurgical service as part of standard of care

Exclusion Criteria:

* Patients older than 21 years of age
* Do not have a Strata CSF shunt valve
* Not patients of the All Children's Hospital neurosurgical service

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients 21 years of age and younger, with Strata valve CSF shunts, who are being evaluated by the All Children's Hospital (ACH) neurosurgical service as part of standard of care, will be eligible for participation during the three-year enrollment period. Each time an eligible patient has contact with the neurosurgical service their valve will be checked for possible inadvertent reprogramming in the outpatient facilities, emergency department, and inpatient setting. Patients will only have their valves checked as part of this study once during each encounter. Only patients who were evaluated by the neurosurgical service and returned to their normal environment more than seven days prior to their current encounter will be eligible to have their valves rechecked as part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Tuite, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Single Ecounter Assessment: Pediatric patients with adjustable cerebral spinal fluid shunt valves were assessed at "single" encounters when scheduled for an MRI. Assessment included questionnaires that assessed multiple variables that have been previously associated with inadvertent reprogramming, including proximity to magnets, iPads and cell phones. Valve settings were assessed before and after the MRI and data collected regarding history, clinical and imaging findings.
Period: Overall Study
Arm/Group | Observational Single Ecounter Assessment
Started | 95 (114 encounter assessments were completed on 95 participants over 15 months)
Completed | 95
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: encounters
Groups:
- Observational Single Encounter Assessment: Pediatric patients with adjustable cerebral spinal fluid shunt valves were assessed at "single" encounters when scheduled for an MRI. Assessment included questionnaires that assessed multiple variables that have been previously associated with inadvertent reprogramming, including proximity to magnets, iPads and cell phones. Valve settings were assessed before and after the MRI and data collected regarding history, clinical and imaging findings.
Arm/Group | Observational Single Encounter Assessment
Number analyzed (Participants) | 95
Number analyzed (encounters) | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 88
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Encounters With Inadvertent Reprogramming of Strata CSF Shunt Valves.
Description: Assessed by checking the valves at routine follow-up visits, in patient hospitalizations and prior to MRI imaging. The frequency will be calculated by the number of encounters/visits during which an assessed valve was inadvertently reprogrammed divided by the total number of encounters/visits in the trial. Here, we report the number of encounters/visits during which valves were inadvertently reprogrammed.
Time Frame: 14 months
Measure: Count of Units; unit: Encounters
Units Other Than Participants: Encounters
Groups:
- Observational Single Ecounter Assessment: Pediatric patients with adjustable cerebral spinal fluid shunt valves were assessed at "single" encounters when scheduled for an MRI. Assessment included questionnaires that assessed multiple variables that have been previously associated with inadvertent reprogramming, including proximity to magnets, iPads and cell phones. Valve settings were assessed before and after the MRI and data collected regarding history, clinical and imaging findidngs.
Arm/Group | Observational Single Ecounter Assessment
Number analyzed (Participants) | 95
Number analyzed (Encounters) | 114
Encounters | 15

2. Secondary Outcome: Number of Encounters/Visits With or Without Valve Changes Due to MRI Field Strengths.
Description: Shunt valve settings were assessed before and after MRI studies using the 1.5 Tesla (T), 3 Tesla (T) or other MRI field strengths for any valve setting changes.
Time Frame: 14 months
Population: Data collected from 91 encounters who underwent MRI either on the 1.5 T or the 3 T as part of their visit
Measure: Count of Units; unit: encounters
Units Other Than Participants: encounters
Arm/Group | Observational Single Ecounter Assessment
Number analyzed (Participants) | 95
Number analyzed (encounters) | 91
encounters
  1.5 T MRI valve changes: valve changes | 76
  1.5 T MRI valve changes: no valve change | 15
  3T MRI valve changes: valve changes | 78
  3T MRI valve changes: no valve change | 13

3. Secondary Outcome: Number of Encounters With Increased Signs, Symptoms and Radiographic Changes Suggestive of Shunt Malfunction in Participants With Inadvertent Reprogramming of the Strata Valve Compared to Those Without Inadvertent Reprogramming.
Description: Increased Signs, Symptoms and Radiographic Changes Suggestive of Shunt Malfunction in Participants With Inadvertent Reprogramming of the Strata Valve Compared to Those Without Inadvertent Reprogramming Assessment will be made using a family questionnaire and data sheet from clinical evaluation.
Time Frame: 14 months
Population: Data collected from the 15 participants with inadvertent reprogramming.
Measure: Number; unit: encounters - signs of shunt malfunction
Units Other Than Participants: encounters with reprogramming
Arm/Group | Observational Single Ecounter Assessment
Number analyzed (Participants) | 15
Number analyzed (encounters with reprogramming) | 15
encounters - signs of shunt malfunction | 7

4. Secondary Outcome: Number of Encounters of Inadvertent Reprogramming With Exposure to Household Devices With Electromagnetic Charge.
Description: Here we report the number of encounter/visits during which valves were inadvertently reprogrammed due to household devices with electromagnetic charge.
Time Frame: 14 months
Measure: Count of Units; unit: encounters
Units Other Than Participants: encounters
Arm/Group | Observational Single Ecounter Assessment
Number analyzed (Participants) | 95
Number analyzed (encounters) | 114
encounters | 15

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Observational Single Ecounter Assessment
All-Cause Mortality (participants affected / at risk) | 1/95
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT02737163/Prot_SAP_000.pdf